Title of study: Effectiveness of microdosed GLP-1 in improving health, quality of life, and longevity measures

NCT number: Not yet assigned

Date of document: August 28, 2024



## Informed Consent Form

Title of Study: Effectiveness of microdosed GLP-1 in improving health, quality of life, and longevity measures

Principal Investigator: Sajad Zalzala

Address: 835 Mason St, Ste A250, Dearborn, MI 48126

Tel: (313) 355-8657 Fax: (888) 655-7536

Email: doctor@agelessrx.com

Sponsor: AgelessRx, Inc.

Address: 2370 E Stadium Blvd #2049 Ann Arbor, MI 48104

Tel:650-503-9990 Fax: 650-729-0869

Email: info@agelessrx.com

Site: This is a decentralized trial. Participants can be located in any of the 50 states

of the USA. All participation will be via

telemedicine using the AgelessRx website (agelessrx.com).

Purpose of the Study: I understand that the purpose of this study is to evaluate the effectiveness of microdosed semaglutide in improving health, quality of life, and longevity.

Participation: I understand that participation in this study will last approximately 6 months. During this period, I will be asked to start taking low doses of a semaglutide therapy, undergo regular health and weight assessments, and adhere to prescribed interventions.

Eligibility: I understand that my eligibility for this study has been assessed following the completion of the informed consent form. This study welcomes participants regardless of ethnicity, gender, socioeconomic status, educational status, sexual preference, religious preference, or political views.

Possible Benefits: I understand that there is no guarantee of personal benefit from participating in this study. The study aims to contribute valuable data to the field of weight management post-semaglutide therapy.

Possible Risks: I understand that participating in this study may involve risks, including but not limited to gastrointestinal discomfort, changes in mood, and other side effects associated with the alternative therapies.

Confidentiality: I understand that my health information will be stored in a secure database and will be accessible only to the study team. Personal information will be closely protected, and I will not be identifiable in any publication resulting from this study.

Costs: I understand that there are no costs required for me to participate in this study. All related expenses will be covered by the sponsor.

Withdrawal: I understand that I am free to withdraw from the study at any time without penalty.

Protocol Number: ALRx-010 Approval Date: August 28, 2024 Approval Number:

IRCM-2024-411 Continuing Review Date: September 24, 2025

## agelessrx

Data Sharing: I understand that de-identified data from this study may be shared with the wider research community to advance science and health, with assurances made to protect my privacy to the best of the sponsor's ability.

Future Use of Data: I understand that de-identified information may be used for future research without additional consent.

Contacting the Research Team: I understand that I have the right to ask any questions and express any concerns by contacting the research team directly at Research@agelessrx.com or (650) 272-3169.

Should I wish to contact an impartial third party not associated with this study, I may contact James P. Faber, secretary of the Institutional Review Board (IRB) of the Institute of Regenerative and Cellular Medicine (IRCM), which reviewed this study for ethical compliance: jpfaber@ircm.org or (786) 271-2156.

By signing below, I confirm that I have read and understood the information provided, have had the opportunity to ask questions, and agree to participate in this study.

Participant Signature: Date: Principal Investigator Signature: